CLINICAL TRIAL: NCT02735538
Title: Transcription Factor Runx2 in Necrotic Femoral Head Tissue: Study Protocol for a Retrospective Non-randomized, Parallel-controlled Clinical Trial
Brief Title: Transcription Factor Runx2 in Necrotic Femoral Head Tissue
Status: Completed | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Liqing Yang, Vice President, Shengjing Hospital
Other Study IDs: ShengjingH_LQYang
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Osteonecrosis of Femoral Head
MeSH Terms: conditions — Femur Head Necrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- osteonecrosis of femoral head group: The patients with osteonecrosis of femoral head undergo total hip replacement. Femoral head specimens will be collected and ex vivo specimens numbered. Using RT-PCR, Runx2, BMP-2, BMP-7 and osteoprotegerin, mRNA expression levels will be quantitatively analyzed. Osteocalcin immunoreactivity will be detected using immunohistochemical staining.
  Interventions: Procedure: osteonecrosis of femoral head group
- osteoarthritis group: The patients with osteoarthritis will undergo total hip replacement. Femoral head specimens will be collected and ex vivo specimens numbered. Using RT-PCR, Runx2, BMP-2, BMP-7 and osteoprotegerin, mRNA expression levels will be quantitatively analyzed. Osteocalcin immunoreactivity will be detected using immunohistochemical staining.
  Interventions: Procedure: osteoarthritis group

INTERVENTIONS:
Procedure: osteonecrosis of femoral head group — The patients with osteonecrosis of femoral head will undergo total hip replacement.
  Groups: osteonecrosis of femoral head group
Procedure: osteoarthritis group — The patients with osteoarthritis will undergo total hip replacement.
  Groups: osteoarthritis group

SUMMARY:
The trial detected mRNA expression of several bone repair-related genes, including Runx2, in the femoral head and neck of patients with osteonecrosis of femoral head (ONFH) . Runx2 expression was compared with that of identical tissue from osteoarthritis patients to identify expression in necrotic femoral head tissue, which will help clarify the role and possible clinical significance of Runx2 in femoral head necrosis, bone repair and reconstruction.

DETAILED DESCRIPTION:
Osteonecrosis of the femoral head (ONFH) is a destructive degenerative disease that can develop into subchondral and articular facet cartilage collapse. Among proposed pathological mechanisms underlying ONFH, much attention has been paid to the theory of increased intraosseous pressure. The core of this theory is an unbalance in osteoblast and adipocyte differentiation of bone marrow mesenchymal stem cells (BM-MSCs). The occurrence and development of osteonecrosis has been related to abnormal metabolism and differentiation of BM-MSCs. Normal adult BM-MSCs can differentiate into adipocytes and osteoblasts to maintain normal physical status. In response to exogenous stimuli (for example, use of exogenous hormones or alcohol), the bone marrow microenvironment changes to allow more BM-MSCs to differentiate into adipocytes, leading to increased bone marrow cavity pressure, thereby inducing ischemic ONFH.

Overexpression of Runx2, an osteoblast-specific transcription factor, can increase osteoblast differentiation of BM-MSCs, thereby strengthening the effects of BM-MSC transplantation to repair bone defects and necrosis. By controlling expression of osteocalcin, an osteoblast-specific gene, Runx2 also controls osteoblast differentiation and functioning. Osteocalcin, a common indicator used to evaluate bone formation and conversion rate, is a bone metabolism-regulating factor generated and secreted by osteoblasts; thus, it is considered to be a good marker for bone functioning. In a previous study by Chen et al., seven patients with glucocorticoid-induced ONFH at Association Research Circulation Osseous (ARCO) Stage IV were included as an experimental group and seven patients with femoral neck fracture served as a control group. Immunohistochemical staining and quantitative polymerase chain reaction (PCR) were used to detect osteocalcin immunoreactivity and Runx2 expression in femoral head and neck tissue. They found that glucocorticoid-induced ONFH is likely closely related to osteocalcin.

ONFH results from an interruption of the blood supply to the femoral head or injury-caused death of chondrocytes and bone marrow components. During subsequent repair processes, bone morphogenetic proteins (BMPs) not only stimulate BM-MSCs to differentiate into osteoblasts, but also promote osteoblast growth; BMP-2 is the key factor regulating bone tissue formation.

Sclerotin loss after ONFH is closely related to an unbalance in osteoclast activity and differentiation. Osteoprotegerin can inhibit bone absorption of mature osteoblasts and induce apoptosis of osteoblasts. Osteoprotegerin and its ligand system have been confirmed as key factors regulating osteoblast formation and differentiation, while bone absorption plays an important role in the pathogenesis and treatment of osteoporosis, osteoarthritis and bone tumors.

To the best of our knowledge, there have been no controlled clinical trials examining BMP, osteocalcin, osteoprotegerin or, in particular, Runx2 messenger RNA (mRNA) expression in femoral head tissue of patients with ONFH at Ficat Stage III-IV and osteoarthritis. In this non-randomized, parallel-controlled trial, we will use real-time PCR (RT-PCR) to detect Runx2, BMP-2, BMP-7 and osteoprotegerin mRNA expression in femoral head tissue from patients with ONFH at Ficat Stage III-IV. Simultaneously, we will detect osteocalcin immunoreactivity using an immunohistochemical staining method, and compare with osteoarthritis patients for the purpose of clarifying mechanisms of these factors in bone reconstruction post-ONFH.

Data collection, management, analysis and open access Data collection: According to the trial design, a table will be formulated for data collection. Collected data will be input into an electronic database by professional staff using a double-data entry strategy.

Data management: Information accuracy will be checked when all recruited patients are followed up. The database will be locked by the researcher in charge and will not be altered. All information relating to this trial will be preserved by Shengjing Hospital of China Medical University, China.

Data analysis: The electronic database will be fully disclosed to a professional statistician for statistical analysis.

Data open access: Published data will be available at www.figshare.com. Statistical analysis Statistical analysis will be performed by a professional statistician (blinded to grouping) using SPSS 19.0 software. If Runx2, BMP-2, BMP-7 and osteoprotegerin mRNA expression, as well as osteocalcin immunoreactivity in the femoral head and neck of patients with ONFH and osteoarthritis, are normally distributed, a two-sample t-test will be used to compare differences between groups. If, however, these data are not normally distributed, a Mann-Whitney U test will be used. A level of P < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as ONFH at Ficat Stage III-IV by anteroposterior and lateral X- ray and/or computed tomography (CT) images
* Diagnosed with hip joint osteoarthritis by laboratory examinations and X-ray images
* Subjected to total hip replacement for the first time
* Able to tolerate anesthesia and surgery
* Provide informed consent regarding the benefits and risks of participation in the trial

Exclusion Criteria:

* Complicated by severe primary cardiovascular disease, hepatic and/or renal inadequacy, or hematopoietic system disorders
* Pregnant or lactating woman
* With blood coagulation disorder
* With a history of epilepsy or mental disorder
* Have participated in other clinical trials within 30 days prior to recruitment
* Are taking part in other clinical trials
* Cannot manage him/herself or have poor self-control ability
* Human immunodeficiency virus (HIV)-positive or hepatitis virus-positive
* Active systemic or local infection
* Poor tolerance to total hip replacement

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifteen patients with ONFH at Ficat Stage III¬-IV and 15 patients with osteoarthritis will undergo total hip replacement. Femoral head specimens will be collected and ex vivo specimens numbered. Using RT-PCR, Runx2, BMP-2, BMP-7 and osteoprotegerin, mRNA expression levels will be quantitatively analyzed. Osteocalcin immunoreactivity will be detected using immunohistochemical staining. Professional staff, blinded to grouping, will perform outcome index detection and statistical analysis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Runx2 mRNA expression in femoral head and neck tissue | During surgery
  Runx2, a primary transcription factor controlling osteoblast commitment and differentiation, can be considered an osteoblast phenotype marker.

SECONDARY OUTCOMES:
bone morphogenetic protein-2(BMP-2) | During surgery
bone morphogenetic protein-7(BMP-7) | During surgery
osteoprotegerin | During surgery
osteocalcin immunoreactivity | During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Liqing Yang, M.D., Principal Investigator — Shengjing Hospital of China Medical University, China

IPD SHARING:
Plan to Share IPD: Undecided